CLINICAL TRIAL: NCT03034083
Title: Elevate: Taking Your Relationship to the Next Level
Brief Title: An Evaluation of Healthy Marriage and Relationship Education Program: Elevate
Status: Withdrawn | Type: Observational
Why Stopped: No subjects recruited
Sponsor: University of Georgia (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, Karen M. DeMeester, Public Service Assistant, University of Georgia
Other Study IDs: 90FM0081
Record Dates: First submitted 2017-01-19; First posted 2017-01-27 (Estimated); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Family Relations
Keywords: healthy marriage; healthy relationships; parenting; healthy marriage and relationship education

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Couples Elevate Weekly Series: Participants in a couple relationship receive needs assessment and 8 hours of classes over a 4-week period in healthy couple functioning behaviors, relationship quality/stability, and parenting skills.
  Interventions: Behavioral: Elevate
- Foster Parents Elevate Weekend Intensive: Foster parent participants receive 8 hours of classes over a weekend in healthy couple functioning behaviors, relationship quality/stability, and parenting skills.

INTERVENTIONS:
Behavioral: Elevate — Study participants receive needs assessment and 8 hours of classes over a 4-week period in healthy couple functioning behaviors, relationship quality/stability, and parenting skills.
  Groups: Couples Elevate Weekly Series

SUMMARY:
The purpose of this study is to determine whether the healthy marriage and relationship education program Elevate: Taking Your Relationship to the Next Level results in improved couple, parenting, and co-parenting behaviors that lead to reduced child abuse/neglect potential.

DETAILED DESCRIPTION:
The descriptive study is based on the theory that couples can learn skills through participating in the Elevate curriculum that will help them function better as a couple resulting in improved relationship quality/stability, improved co-parenting skills, improved financial management, and reduced financial stress. As a result of improved relationship skills and better management of stress, couples will then provide more supportive, safe, and stable family environments for children.

Individuals who are eligible (biological and foster parents of children 0-18) and agree to participate in the study will complete surveys at three time points--before participating in Elevate, 4-6 weeks after participating, and 8-10 months after participating in Elevate. The surveys include items related to couple functioning behaviors, relationship quality/stability, parenting/co-parenting skills, and financial management and distress.

ELIGIBILITY:
Inclusion Criteria:

Biological parents of children 0-18 Parents must be in a committed couple relationship

Exclusion Criteria:

Incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is biological and foster parents of children ages 0-18.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Elevate Pre-post program survey subscale measuring change in couple functioning and stability | Time points 4-6 weeks prior to participation in Elevate, 4-6 week after participation, and 8-10 months after participation.
  Study participant responses on Elevate pre-post survey subscale measuring change in couple functioning behaviors, including communication, conflict resolution, commitment, and supportive behaviors will be compared at three time points.

SECONDARY OUTCOMES:
Elevate Pre-post survey subscale measuring change in parenting skills | Time points 4-6 weeks prior to participation in Elevate, 4-6 week after participation, and 8-10 months after participation
  Study participant responses on Elevate pre-post survey subscale measuring change in parenting skill level, including interactions with children, co-parenting approaches, and beliefs about appropriate parenting behaviors, will be compared at three time points.

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Futris, Ph.D., Principal Investigator — University of Georgia
Locations (1):
- University of Georgia, Athens, Georgia, United States

IPD SHARING:
Plan to Share IPD: No